CLINICAL TRIAL: NCT01147315
Title: 10 Patients Bicentric Prospective Study of Hybrid Bone Substitution With Calcium-phosphate Ceramic Biomaterial and Autologous Bone Marrow for Mandibular Osteoradionecrosis (ORN) Treatment
Brief Title: ORN Study: Curative Treatment of Osteoradionecrosis (ORN) With Hybrid Bone Substitution
Acronym: ORN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRD/08/10-H
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2017-05

CONDITIONS: Mandible; Osteoradionecrosis
Keywords: mandibular osteoradionecrosis; hybrid bone substitution; calcium-phosphate ceramic biomaterial; autologous bone marrow
MeSH Terms: conditions — Osteoradionecrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hybrid bone substitution (Experimental): Hybrid bone substitution with calcium-phosphate ceramic biomaterial and autologous bone marrow
  Interventions: Procedure: Hybrid bone substitution

INTERVENTIONS:
Procedure: Hybrid bone substitution — The patient will be treated by hybrid bone substitution with calcium-phosphate ceramic biomaterial and autologous bone marrow after necrosis exeresis

SUMMARY:
The main objective of the study is the cure of osteoradionecrosis (ORN) at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (between 18 and 75 years) affiliated with an appropriate social security system, diagnosed as suffering from symptomatic ORN, radiologically confirmed, for which surgery is indicated
* Presence maximum of 2 outbreaks of ORN
* Oncological remission of the original tumor site for 1 year and for 3 years if the ORN is in the contact or close to the initial tumoral site
* ECOG performance status 0, 1 or 2
* ORN symptomatic accessible to the conservation of at least one cortical mandibular basilar
* Signed informed consent

Exclusion Criteria:

* Oncological treatment
* Haematologic background
* Current bone necrosis consecutive or concurrent to taking bisphosphonates
* Extension of ORN does not allow the retention of a mandibular rod (bicortical form)
* Presence of fracture complicating ORN
* Bisphosphonates during the last year
* Contraindications to the removal of iliac or sternum bone marrow
* Contraindication for general anesthesia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-11-18; Primary Completion 2016-11-16 (Actual); Study Completion 2016-11-16 (Actual)

PRIMARY OUTCOMES:
The cure of ORN | 12 months

SECONDARY OUTCOMES:
Evaluation of post operative pain at mandibular and bone marrow sampling site
Quality of life
Possibility of secondary dental prosthetic devices
CT semiology description of the treated area
Bone regeneration
  Bone regeneration: kinetics of formation of new bone and biomaterial resorption
Number of hospital days
Safety of hybrid bone substitution

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Malard, Pr, Principal Investigator — Nantes University Hospital
Locations (2):
- France (2):
  - Nantes University Hospital, Nantes
  - Rennes University Hospital, Rennes